CLINICAL TRIAL: NCT03018990
Title: Alcohol Challenge On Liver and Gut Measured by Liver Vein Catheterization. A Pathophysiological Intervention Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mads Israelsen, MD,clinical research assistant, PhD-student, Odense University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: S-20160083
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Liver Fibroses; Alcohol-Induced Disorders
MeSH Terms: conditions — Liver Cirrhosis; Alcohol-Induced Disorders | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alcoholic liver fibrosis (Active Comparator)
  Interventions: Other: Ethanol
- Non-alcoholic steatohepatitis (Active Comparator)
  Interventions: Other: Ethanol
- Healthy control (Active Comparator)
  Interventions: Other: Ethanol

INTERVENTIONS:
Other: Ethanol — 1 milliliter per kilogram body weight adjusted for elevated body mass index

SUMMARY:
To investigate the effects of acute alcohol challenge on the gut and liver axis.

DETAILED DESCRIPTION:
To study the role of acute alcohol challenge on the intestine permeability and inflow of bacterial products to the liver in participants with alcoholic liver disease, non-alcoholic steatohepatitis and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Alcoholic liver fibrosis, non-alcoholic steatohepatitis or liver-healthy individuals

And all of following:

* Bodymass > 50 kg
* Able to be fasting and abstinent on the day of intervention
* international ratio <1.5 and platelets >100 x 10^9, 7 days before the intervention day
* Informed consent

Exclusion Criteria:

* Antibiotics during the last 4 weeks
* Total alcohol abstinence
* Desire of total alcohol abstinence
* Other causes of liver disease suspected (viral, autoimmune, haemochromatosis, Wilsons diseases, alfa 1 antitrypsin deficiency or drug induced)
* Cirrhosis
* Insulin dependent diabetes mellitus
* Incapable to follow the protocol instructions
* Pregnancy
* Primary or secondary liver cancer
* Severe comorbidity
* Allergic to the contrast media iohexol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
changes in concentrations of bacterial products in the liver vein | Within 24 hours

SECONDARY OUTCOMES:
changes in concentrations of bacterial products in the peripheral vein system | Within 24 hours
changes in the gut microbiome | Within 24 hours
changes in the liver metabolome, transcriptome and proteome | Within 24 hours
changes in serum-ethanol, plasma-glucose and liver biomarkers in the liver vein compared to the peripheral vein system | Within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Aleksander Krag, MD, PhD, Principal Investigator — Professor, department of gastroenterology and hepatology, Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Fyn, Denmark

REFERENCES:
- [Derived] Stankevic E, Israelsen M, Juel HB, Madsen AL, Angquist L, Aldiss PSJ, Torp N, Johansen S, Hansen CD, Hansen JK, Thorhauge KH, Lindvig KP, Madsen BS, Sulek K, Legido-Quigley C, Thiele MS, Krag A, Hansen T. Binge drinking episode causes acute, specific alterations in systemic and hepatic inflammation-related markers. Liver Int. 2023 Dec;43(12):2680-2691. doi: 10.1111/liv.15692. Epub 2023 Aug 17. PMID 37592403
- [Derived] Israelsen M, Kim M, Suvitaival T, Madsen BS, Hansen CD, Torp N, Trost K, Thiele M, Hansen T, Legido-Quigley C, Krag A; MicrobLiver Consortium. Comprehensive lipidomics reveals phenotypic differences in hepatic lipid turnover in ALD and NAFLD during alcohol intoxication. JHEP Rep. 2021 Jun 29;3(5):100325. doi: 10.1016/j.jhepr.2021.100325. eCollection 2021 Oct. PMID 34401690